CLINICAL TRIAL: NCT06188520
Title: A Phase I/IIa, First-in-human, Open-label, Dose Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of AZD8421 Alone or in Combination in Participants With Selected Advanced or Metastatic Solid Tumors
Brief Title: A First-in-human Dose Escalation and Expansion Study to Evaluate the Safety, and Tolerability of AZD8421 Alone or in Combination in Participants With Selected Advanced or Metastatic Solid Tumors
Acronym: CYCAD-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8470C00001
Record Dates: First submitted 2023-12-01; First posted 2024-01-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: ER+ HER2- Advanced Breast Cancer; High-grade Serous Ovarian Cancer (HGSOC)
MeSH Terms: interventions — AZD9833; ribociclib; palbociclib; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1 (Experimental): AZD8421 monotherapy
  Interventions: Drug: AZD8421
- Module 2A (Experimental): AZD8421 with camizestrant and CDK4/6 inhibitor
  Interventions: Drug: AZD8421; Drug: Camizestrant; Drug: Ribociclib; Drug: Palbociclib; Drug: Abemaciclib

INTERVENTIONS:
Drug: AZD8421 — CDK2 inhibitor
Drug: Camizestrant — SERD
  Other Names: AZD9833
  Arms: Module 2A
Drug: Ribociclib — CDK4/6 inhibitor
  Other Names: Kisqali
  Arms: Module 2A
Drug: Palbociclib — CDK4/6 inhibitor
  Other Names: Ibrance
  Arms: Module 2A
Drug: Abemaciclib — CDK4/6 inhibitor
  Other Names: Verzenios
  Arms: Module 2A

SUMMARY:
This study is designed to evaluate AZD8421 alone and in combination with selected targeted anti-cancer drugs in patients with ER+HER2- advanced breast cancer, and patients with metastatic high-grade serious ovarian cancer.

DETAILED DESCRIPTION:
This is a first in-human study of AZD8421 administered to participants with advanced or metastatic solid tumors. The study will evaluate the safety, tolerability, preliminary efficacy, pharmacokinetics, and pharmacodynamics of AZD8421 alone and in combination with selected targeted anti-cancer drugs.

AZD8421 monotherapy (M1) will evaluate the safety, tolerability and pharmacokinetics of AZD8421 as monotherapy to identify a recommended Phase II dose (RP2D) in participants with ER+ HER2- advanced breast cancer previously treated with a CDK4/6i (Parts A and B) and participants with metastatic high-grade serous ovarian cancer previously treated with a platinum-based chemotherapy in the metastatic setting (Part B).

AZD8421 combination therapy (M2) will evaluate the safety, tolerability, and pharmacokinetics of different formulations of AZD8421 in combination with a CDK4/6 inhibitor (one or more of abemaciclib, ribociclib and palbociclib) and camizestrant (next generation oral SERD; referred to throughout as 'camizestrant') in participants with ER+ HER2- advanced breast cancer previously treated with a CDK4/6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Female participants only, aged 18 or above
* Participants with advanced solid tumors must have received prior adequate therapy in accordance with local practice for their tumor type and stage of disease, or, in the opinion of the Investigator, a clinical study is the best option for their next treatment based on response to and/or tolerability of prior therapy.
* Metastatic or locoregionally recurrent disease and radiological or objective evidence of progression on or after the last systemic therapy prior to starting IMP.
* ECOG/WHO performance status 0 to 1, and a minimum life expectancy of 12 weeks.
* At least one lesion that is measurable and/or non-measurable, as per RECIST v1.1 and that can be accurately assessed at baseline and is suitable for repeated assessment.

Exclusion Criteria:

* Intervention with any of the following:
* Any cytotoxic chemotherapy, investigational agents, or other anti-cancer drugs for the treatment of advanced cancer from a previous treatment regimen or clinical study within 14 days or 5 half-lives (whichever is shorter) of the first dose of IMP (21 days for myelosuppressive therapies) other than GnRHa (eg, goserelin) and bone-stabilizing agents (eg, zoledronic acid, denosumab).
* Any prescription or non-prescription drugs or other products, including herbal products, known to be moderate or strong inhibitors/inducers of CYP3A4/5 which cannot be discontinued prior to first dose of IMP and withheld throughout the study until 2 weeks after the last dose of study drug.
* Drugs that have a known risk of Torsades de Pointes.
* Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of IMP.
* Major surgical procedure or significant traumatic injury, within 4 weeks of the first dose of IMP, or an anticipated need for major surgery and/or any surgery requiring general anesthesia during the study.
* Any unresolved toxicities of Grade ≥ 2 from prior anti-cancer therapy (with the exception of alopecia). Participants with stable ≤ Grade 2 neuropathy are eligible.
* Presence of life-threatening metastatic visceral disease, as judged by the Investigator, uncontrolled CNS metastatic disease. Participants with spinal cord compression and/or brain metastases may be enrolled if definitively treated (eg, surgery or radiotherapy) and stable off steroids for at least 4 weeks prior to start of IMP.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, or eg, infection requiring IV antibiotic therapy, or active infection including hepatitis B, hepatitis C, and HIV (active viral infection is defined as requiring antiviral therapy; screening for chronic conditions is not required).
* Any of the following cardiac criteria:
* Mean resting QTcF > 470 msec obtained from a triplicate ECG
* Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (eg, complete left bundle branch block, second- and third-degree heart block), or clinically significant sinus pause. Participants with controlled atrial fibrillation can be enrolled.
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as symptomatic heart failure, hypokalemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death at < 40 years of age. Hypertrophic cardiomyopathy and clinically significant stenotic valve disease.
* LVEF < 50%, and/or experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, unstable angina pectoris, congestive heart failure NYHA Grade ≥ 2, cerebrovascular accident, or transient ischemic attack.
* Uncontrolled hypertension.
* Inadequate bone marrow reserve or organ function as demonstrated by relevant laboratory values:
* Refractory nausea and vomiting, uncontrolled chronic gastrointestinal diseases, or previous significant bowel resection that would preclude adequate absorption of IMP(s).
* History of hypersensitivity to active or inactive excipients of AZD8421 or drugs with a similar chemical structure or class to AZD8421.
* Previous treatment with AZD8421 or with any CDK2-selective inhibitor, or protein kinase membrane-associated tyrosine- and threonine-specific cdc2-inhibitory kinase 1 (PKMYT1) inhibitor, or WEE1 inhibitor.
* Currently pregnant (confirmed with positive pregnancy test), breast feeding, or planning to become pregnant. Participants of childbearing potential must agree to use one highly effective contraceptive measure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) as defined in the protocol. | From start of treatment until the end of DLT period, assessed up to 28 days.
  Percentage of participants with incidence of DLTs.
Incidence of AEs/SAEs | From start of treatment until the end of safety follow-up, approximately 18 months.
  Percentage of participants with incidence of AEs/SAEs.
Clinically significant changes from baseline in clinical laboratory parameters, vital signs and ECGs. | From start of treatment until the end of safety follow-up, approximately 18 months.
  Percentage of participants with clinically significant changes from baseline in clinical laboratory parameters, vital signs and ECGs.
Discontinuation of AZD8421 due to toxicity | From start of treatment until the end of safety follow-up, approximately 18 months.
  Percentage of participants that have discontinued AZD8421 due to toxicity.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 8 weeks from start of treatment until end of treatment or objective disease progression, approximately 18 months.
  The percentage of participants with a confirmed Complete Response (CR) or Partial Response (PR), according to RECIST v1.1, that occur prior to disease progression and/or initiation of subsequent anti-cancer therapy.
Duration of Response (DoR) | 8 weeks from start of treatment until end of treatment or objective disease progression, approximately 18 months.
  The time from the date of first documented objective response (which is subsequently confirmed) until date of first documented disease progression or death (by any cause in the absence of disease progression).
Disease control rate (DCR) | 24 weeks after the start of treatment.
  The percentage of participants who have a best objective response of confirmed CR or PR or who have SD for at least 23 weeks after start of treatment.
Percentage change in tumor size | From start of treatment through to EOT, progressive disease, death (in the absence of progression), start of subsequent anti-cancer therapy, whichever occurs first, approximately 18 months.
  The largest decrease (or smallest increase) in tumor size from baseline for a participant, using RECIST v1.1 assessments
Progression Free Survival (PFS) | From start of treatment through to progressive disease, death (in the absence of progression), EOT (last evaluable disease assessment), whichever occurs first, approximately 18 months.
  Progression-free survival is defined as the time from the start of treatment until the date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the participant withdraws from therapy or receives another anti-cancer therapy prior to progression.
PK of AZD8421 (Cmax) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After single dose; Cmax; to measure maximum plasma concentration after oral administration.
PK of AZD8421 (Tmax) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After single dose; Tmax; to measure time to reach maximum plasma concentration.
PK of AZD8421 (AUCinf) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After single dose; AUCinf; to measure the area under the plasma concentration-time curve from time 0 to infinity.
PK of AZD8421 (AUClast) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After single dose; AUClast; to measure area under the plasma concentration-time curve from time zero to last PK sample.
PK of AZD8421 (T1/2λZ) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After single dose; T1/2λZ; to measure the terminal elimination half-life.
PK of AZD8421 (CL/F) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After single dose; CL/F; to measure apparent clearance after oral administration.
PK of AZD8421 (Cssmax) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After multiple doses; Cssmax; to measure maximum concentration after oral administration at steady state.
PK of AZD8421 (Tssmax) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After multiple doses; Tssmax; to measure time it takes to achieve maximum plasma concentration at steady state.
PK of AZD8421 (ARCmax) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After multiple doses; ARCmax; to measure accumulation ratio of Cmax.
PK of AZD8421 (AUCsslast) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After multiple doses; AUCsslast; to measure the area under plasma-concentration time curve from time zero to last PK sample at steady state.
PK of AZD8421 (T1/2λssz) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After multiple doses; T1/2λssz; to measure terminal elimination half-life at steady state.
PK of AZD8421 (CLss/F) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after single and multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After multiple doses; CLss/F; to measure apparent oral clearance at steady state.
PK of AZD8421, camizestrant, and CDK4/6i (Cmax) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After single dose: Cmax; to measure maximum plasma concentration after oral administration.
PK of AZD8421, camizestrant, and CDK4/6i (Tmax) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After single dose: Tmax; to measure the time it takes to achieve maximum plasma concentration after oral administration.
PK of AZD8421, camizestrant, and CDK4/6i (AUCinf) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After single dose: AUCinf; to measure area under plasma concentration-time curve from time zero to infinity.
PK of AZD8421, camizestrant, and CDK4/6i (T1/2λ) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After single dose: T1/2λZ; to measure terminal elimination half-life.
PK of AZD8421, camizestrant, and CDK4/6i (CL/F) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After single dose: CL/F; to measure apparent clearance after oral administration.
PK of AZD8421, camizestrant, and CDK4/6i (Cssmax) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After multiple doses: Cssmax; to measure the maximum plasma concentration after oral administration at steady state.
PK of AZD8421, camizestrant, and CDK4/6i (Tssmax) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After multiple doses: Tssmax; to measure time it takes to achieve maximum plasma concentration after oral administration at steady state.
PK of AZD8421, camizestrant, and CDK4/6i (AUC0-tau) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After multiple doses: AUC0-tau; to measure area under plasma-concentration-time curve within dosing interval.
PK of AZD8421, camizestrant, and CDK4/6i (T1/2λssz) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After multiple doses: T1/2λssz; to measure terminal elimination half-life at steady state.
PK of AZD8421, camizestrant, and CDK4/6i (CLss/F) (M2 only) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421, camizestrant and CDK4/6i.
  Evaluate pharmacokinetics profiles of AZD8421, camizestrant, and CDK4/6i when administered in combination.
  For AZD8421 and where possible CDK4/6i and their metabolites, and camizestrant; descriptive statistics of the following PK parameters:
  After multiple doses: CLss/F; to measure apparent clearance after oral administration at steady state.
PD of AZD8421 (M1B only) | Baseline and Cycle 1 Day 15.
  To assess pharmacodynamic activity of AZD8421 monotherapy by assessment of candidate biomarker in baseline and on-treatment tumor and blood samples in participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
PK of AZD8421 (ARAUC) | From start of treatment, at predefined intervals up to Cycle 6, approximately 6 months (each cycle is 28 days) of the administration of AZD8421.
  To characterize the PK profiles and parameters of AZD8421 and its metabolites after monotherapy and also in combination with other anti-cancer drugs after multiple doses when administered to participants with ER+ HER2- metastatic breast cancer and other advanced solid tumors.
  Descriptive statistics of following PK parameters:
  After multiple doses measure accumulation ratio of AUC.
Best Objective Response (BOR) | 8 weeks from start of treatment until end of treatment or objective disease progression, approximately 18 months.
  The best response a participant has had following start of dosing, but prior to starting any subsequent cancer therapy and up to and including date of first documented disease progression, last evaluable assessment or death (by any cause in the absence of disease progression).

CONTACTS AND LOCATIONS:
Overall Officials: Richard Baird, MD, PhD, Study Chair — Cambridge University Hospitals
Locations (13):
- United States (4):
  - Research Site, St Louis, Missouri
  - Research Site, Providence, Rhode Island
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
- Research Site, East Melbourne, Australia
- Research Site, Seoul, South Korea
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Pamplona
  - Research Site, Valencia
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home